CLINICAL TRIAL: NCT01218061
Title: IT-DIAB (Therapeutic Innovation in Type 2 Diabetes) : Prospective Follow-up of a Cohort of Patients With Pre-diabetes Over 10 Years
Brief Title: Therapeutic Innovation in Type 2 DIABetes (IT-DIAB)
Acronym: IT-DIAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROG/09/11
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Pre-diabetes
Keywords: Pre-diabetes; Type 2 diabetes; Biomarkers; Cohort; Diabetes Risk Score
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pre-diabetes screening — The timing of the study is :- Screening of high metabolic risk patients based on a clinical score : Finnish Diabetes Risk Score ≥ 15- if Diabetes Risk Score ≥ 15 or if history of blood glucose between 1.10 and 1.26 g/l (impaired fasting glucose): measuring fasting glycaemia + HbA1C + lipids profile + creatinemia + liver enzymes- if fasting blood glucose between 1.10 and 1.26 g/l (=V0):* OGTT (oral glucose tolerance test) to identify subjects with impaired glucose tolerance (optional)* establishment of a serum bank to identify biomarkers (serum, genomic, proteomic) - to plan for 10 years annual follow-up (V1 to V10) with blood sample (fasting glycemia + HbA1C + lipids profile + creatinemia + liver enzymes + serum bank (not after V5)) Making a total of 11 visits (V0-V10) with 6 blood samples.

SUMMARY:
The main objective of the study is to follow prospectively a cohort of patients with pre-diabetes to understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Subjects with diabetes risk score ≥ 15
* Subjects with impaired fasting glucose: blood glucose ≥ 1.10 g/l and < 1 .26 g/L
* Subjects affiliated with an appropriate social security system

Exclusion Criteria:

* Fasting glycemia ≥ 1.26 g/l
* Fasting glycemia ≤ 1.10 g/l
* Subjects previously treated with oral anti-diabetic: metformin, glitazones, inhibitors of α-glucosidase, sulfonylurea, repaglinide, inhibitors of DPP-IV, GLP-1 R agonists.
* Subjects previously treated with insulin, except gestational diabetes
* Severe coagulation disorders
* Thrombocytopenia < 100 000/mm 3
* Severe psychiatric disorders
* Severe renal insufficiency (creatinine clearance < 30 ml/min)
* Severe hepatic insufficiency (TP < 50%)
* Alcohol abuse (> 30g/j)
* Patient's opposition
* Subject unable to follow the study during the 5 years of follow-up
* Subject exclusion period in a previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The main objective of the study is to understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in this population | 10 years
  The main objective of the study is to follow prospectively a cohort of patients with pre-diabetes to understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in this population

SECONDARY OUTCOMES:
Number of patients with pre-diabetes | 10 years
  To evaluate the prevalence of pre-diabetes in the region of Nantes
HbA1c measurement | 10 years
  To evaluate the role of HbA1C in screening for pre-diabetes and T2D
Number of patients with high Diabetes Risk Score and pre-diabetes | 10 years
  To evaluate the interest of the Diabetes Risk Score in identifying subjects with pre-diabetes in the French population
Number of patients with others cardiovascular risk factors | 10 years
  To evaluate the prevalence of others cardiovascular risk factors associated with pre-diabetes: dyslipidemia, hypertension, metabolic liver disease
Relation between "working hours and conditions" and metabolic disease | 10 years
  To evaluate the impact of working hours and conditions on the prevalence of metabolic diseases (pre-diabetes, dyslipidemia…)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Cariou, Pr, Principal Investigator — University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Rodrigues Oliveira A, Chevalier C, Wargny M, Pakulska V, Caradeuc C, Cloteau C, Letertre MPM, Giraud N, Bertho G, Bigot-Corbel E, Carpentier M, Nouadje G, Coute Y, Le May C, Cariou B, Hadjadj S, Croyal M. Methylglyoxal-Induced Glycation of Plasma Albumin: From Biomarker Discovery to Clinical Use for Prediction of New-Onset Diabetes in Individuals with Prediabetes. Clin Chem. 2025 Jun 3;71(6):688-699. doi: 10.1093/clinchem/hvaf035. PMID 40192447
- [Derived] Croyal M, Wargny M, Chemello K, Chevalier C, Blanchard V, Bigot-Corbel E, Lambert G, Le May C, Hadjadj S, Cariou B. Plasma apolipoprotein concentrations and incident diabetes in subjects with prediabetes. Cardiovasc Diabetol. 2022 Feb 7;21(1):21. doi: 10.1186/s12933-022-01452-5. PMID 35130909
- [Derived] Chavez-Talavera O, Wargny M, Pichelin M, Descat A, Vallez E, Kouach M, Bigot-Corbel E, Joliveau M, Goossens JF, Le May C, Hadjadj S, Hanf R, Tailleux A, Staels B, Cariou B. Bile acids associate with glucose metabolism, but do not predict conversion from impaired fasting glucose to diabetes. Metabolism. 2020 Feb;103:154042. doi: 10.1016/j.metabol.2019.154042. Epub 2019 Nov 27. PMID 31785259
- [Derived] Wargny M, Smati S, Pichelin M, Bigot-Corbel E, Authier C, Dierry V, Zair Y, Jacquin V, Hadjadj S, Boursier J, Cariou B. Fatty liver index is a strong predictor of changes in glycemic status in people with prediabetes: The IT-DIAB study. PLoS One. 2019 Aug 29;14(8):e0221524. doi: 10.1371/journal.pone.0221524. eCollection 2019. PMID 31465427